CLINICAL TRIAL: NCT00251550
Title: Phase I/II Study of LY231514 Plus Cisplatin in Patients With Malignant Pleural Mesothelioma
Brief Title: Study of Pemetrexed Plus Cisplatin in Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5249; H3E-JE-ME01
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Malignant Pleural Mesotherioma
MeSH Terms: interventions — Pemetrexed; Cisplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Cisplatin

SUMMARY:
To investigate efficacy and safety of pemetrexed combined with cisplatin for chemo-naive patients with Malignant Pleural Mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Inapplicable for radical operation
* Not received prior systemic chemotherapy
* Performance status: 0-1

Exclusion Criteria:

* Having a history of sensitivity to platinum agent, folic acid or vitamin B12

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-10; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine the recommended dose of LY231514 and cisplatin combination therapy, Response Rate

SECONDARY OUTCOMES:
Duration of response
Progression free survival
Median survival time
1 year survival rate
Pulmonary function
QOL
Safety
Plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time(UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com